CLINICAL TRIAL: NCT05384249
Title: A Phase 2b Pivotal Study to Evaluate the Efficacy and Safety of Izokibep in Subjects with Non-infectious, Intermediate-, Posterior- or Pan-uveitis
Brief Title: Phase 2b Pivotal Study of Izokibep in Non-infectious, Intermediate-, Posterior- or Pan-uveitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study primary and secondary endpoints did not achieve statistical significance.
Sponsor: ACELYRIN Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21103; 2024-514975-16-00 (EU CTIS Number)
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Uveitis
Keywords: Non-infectious uveitis; Intermediate-uveitis; Posterior-uveitis; Pan-uveitis
MeSH Terms: conditions — Uveitis; Uveitis, Intermediate; Uveitis, Posterior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Placebo subcutaneous once weekly (Placebo Comparator): Participants will receive placebo every week to week 51.
  Interventions: Drug: Placebo
- Group 2: Izokibep subcutaneous once weekly (Experimental): Participants will receive izokibep every week to week 51.
  Interventions: Drug: Izokibep

INTERVENTIONS:
Drug: Izokibep — Biologic: IL-17A inhibitor
  Form: Solution for injection
  Route of administration: Subcutaneous (SC)
  Arms: Group 2: Izokibep subcutaneous once weekly
Drug: Placebo — Form: Solution for injection
  Route of administration: Subcutaneous (SC)
  Arms: Group 1: Placebo subcutaneous once weekly

SUMMARY:
Izokibep is a small protein molecule that acts as a selective, potent inhibitor of interleukin-17A, to which it binds with high affinity. This study investigates izokibep in subjects with active non-infectious, intermediate-, posterior- or pan-uveitis requiring high-dose steroids.

ELIGIBILITY:
Inclusion Criteria:

General

* Subject has provided signed informed consent including consenting to comply with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* 18 years to 75 years of age

Type of Subject and Disease Characteristics

* Subject is diagnosed with non-infectious intermediate-, posterior- or pan-uveitis
* Active disease defined by the presence of at least 1 of the following criteria in at least 1 eye despite treatment with stable doses of corticosteroids for at least 2 weeks prior to day 1:

  * Active, inflammatory, chorioretinal and/or inflammatory retinal vascular lesion by dilated indirect ophthalmoscopy, fundus photography, fluorescein angiography (FA), and Spectral-Domain Optical Coherence Tomography (SD-OCT) to determine whether a lesion is active or inactive (the central reading center assessment using FA, fundus photography and/or SD-OCT is required to confirm eligibility prior to day 1).
  * ≥ 2+ vitreous haze (National Eye Institute [NEI]/Standardization of Uveitis Nomenclature [SUN] criteria) by digital indirect ophthalmoscope and fundus photography (the central reading center assessment using fundus photography is required to confirm eligibility prior to day 1).
* Currently receiving treatment with oral corticosteroids (≥ 7.5 mg/day to ≤ 40 mg/day oral prednisone/prednisolone or corticosteroid equivalent) at a stable dose for at least 2 weeks prior to day 1.

Exclusion Criteria:

Disease-related Medical Conditions

* Subject with isolated anterior uveitis
* Subject with serpiginous choroidopathy
* Subject with confirmed or suspected infectious uveitis
* Subject with corneal or lens opacity that precludes visualization of the fundus or that likely requires cataract surgery during the duration of the study
* Subject with intraocular pressure of ≥ 25 mmHg while on ≥ 2 glaucoma medications or evidence of glaucomatous optic nerve injury
* Subject with severe vitreous haze that precludes visualization of the fundus prior to first dose of study drug
* Subject has a contraindication for mydriatic eye drops OR subject cannot be dilated sufficiently well to permit good fundus visualization
* Subject with best corrected visual acuity (BCVA) < 20 letters (Early Treatment Diabetic Retinopathy Study [ETDRS]) in at least 1 eye prior to first dose of study drug
* Subject with proliferative or severe non-proliferative retinopathy or clinically significant macular edema due to diabetic retinopathy
* Subject with neovascular/wet age-related macular degeneration
* Subject with an abnormality of the vitreo-retinal interface with the potential for macular structural damage independent of the inflammatory process
* Subject with a history of active scleritis ≤ 12 months of first dose of study drug

Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure defined as reaching treatment failure by meeting ≥ 1 of the 4 criteria specified in the protocol in at least 1 eye. | Up to Week 52

SECONDARY OUTCOMES:
Change in best corrected visual acuity (BCVA) from best state achieved | Before Week 10 to Week 24
Change in the National Eye Institute (NEI) Visual Function Questionnarie-25 (VFQ-25) score from best state achieved | Before Week 10 to Week 24
Change in central retinal thickness by Spectral-Domain Optical Coherence Tomography (SD-OCT) | Baseline to Week 10
Change in central retinal thickness by Spectral-Domain Optical Coherence Tomography (SD-OCT) from best state achieved | Week 10 up to Week 52
Proportion of subjects that achieve quiescence | Week 10
Incidence of treatment-emergent adverse events (TEAEs) | Baseline up to Follow-up (Week 65)
Incidence of serious adverse events (SAEs) | Baseline up to Follow-up (Week 65)
Incidence of clinically significant changes in laboratory values | Baseline up to Follow-up (Week 65)
Incidence of clinically significant changes in vital signs | Baseline up to Follow-up (Week 65)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Betah, Study Director — ACELYRIN Inc.
Locations (55):
- United States (32):
  - Clinical Research Site, Phoenix, Arizona
  - Clinical Research Site, Bakersfield, California
  - Clinical Research Site, Beverly Hills, California
  - Clinical Research Site, Los Angeles, California
  - Clinical Research Site, Palo Alto, California
  - Clinical Research Site, Pasadena, California
  - Clinical Research Site, Redlands, California
  - Clinical Research Site, Sacramento, California
  - Clinical Research Site, San Francisco, California
  - Clinical Research Site, Denver, Colorado
  - Clinical Research Site, Clearwater, Florida
  - Clinical Research Site, Marietta, Georgia
  - Clinical Research Site, Oak Park, Illinois
  - Clinical Research Site, Indianapolis, Indiana
  - Clinical Research Site, Hagerstown, Maryland
  - Clinical Research Site, Waltham, Massachusetts
  - Clinical Research Site, Detroit, Michigan
  - Clinical Research Site, Palisades Park, New Jersey
  - Clinical Research Site, New York, New York
  - Clinical Research Site, Winston-Salem, North Carolina
  - Clinical Research Site, Cleveland, Ohio
  - Clinical Research Site, Portland, Oregon
  - Clinical Research Site, Erie, Pennsylvania
  - Clinical Research Site, Pittsburgh, Pennsylvania
  - Clinical Research Site, Charleston, South Carolina
  - Clinical Research Site, Nashville, Tennessee
  - Clinical Research Site, Austin, Texas
  - Clinical Research Site, Bellaire, Texas
  - Clinical Research Site, Houston, Texas
  - Clinical Research Site, Plano, Texas
  - Clinical Research Site, Spokane, Washington
  - Clinical Research Site, Madison, Wisconsin
- Austria (3):
  - Clinical Research Site, Graz
  - Clinical Research Site, Salzburg
  - Clinical Research Site, Vienna
- Czechia (3):
  - Clinical Research Site, Brno
  - Clinical Research Site, Pardubice
  - Clinical Research Site, Prague
- France (3):
  - Clinical Research Site, Lyon
  - Clinical Research Site, Marseille
  - Clinical Research Site, Paris
- Germany (6):
  - Clinical Research Site, Berlin
  - Clinical Research Site, Bonn
  - Clinical Research Site, Hamburg
  - Clinical Research Site, Kiel
  - Clinical Research Site, Leipzig
  - Clinical Research Site, Münster
- Italy (2):
  - Clinical Research Site, Milan
  - Clinical Research Site, Reggio Emilia
- Spain (6):
  - Clinical Research Site, Barcelona
  - Clinical Research Site, Madrid
  - Clinical Research Site (4007), Santiago de Compostela
  - Clinical Research Site (4008), Santiago de Compostela
  - Clinical Research Site, Valencia
  - Clinical Research Site, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided